CLINICAL TRIAL: NCT06614907
Title: A Randomized, Double-blinded, Parallel, Single-dose, PhaseⅠComparative Study to Evaluate the Pharmacokinetics and Safety of QL2108 to Dupixent® in Healthy Chinese Adult Subjects
Brief Title: A PhaseⅠ Comparative Study to Evaluate the Pharmacokinetics of QL2108 to Dupixent®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QL2108-101
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-09

CONDITIONS: Atopic Dermatitis
Keywords: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2108 injection (Experimental): QL2108 injection; 300mg/2.0mL; subcutaneous injection
  Interventions: Drug: QL2108 injection
- Dupixent® (Active Comparator): Dupixent®; 300mg/2.0mL; subcutaneous injection
  Interventions: Drug: Dupixent®

INTERVENTIONS:
Drug: QL2108 injection — 300mg/2.0mL; single dose; prefilled syringe; subcutaneous injection
  Arms: QL2108 injection
Drug: Dupixent® — 300mg/2.0mL; single dose; prefilled syringe; subcutaneous injection
  Arms: Dupixent®

SUMMARY:
It is a randomized, double-blinded, parallel, single-dose, PhaseⅠcomparative study to evaluate the pharmacokinetics and safety of QL2108 to Dupixent® in healthy Chinese adult subjects. A total of 198 healthy subjects are planned to be included and randomized at a ratio of 1:1 to receive single 300mg/2.0ml QL2108 injection or Dupixent®.

DETAILED DESCRIPTION:
The study has a screening period of 28 days. PK blood samples will be collected from subjects to determine the serum concentration of Dupilumab, thus to evaluate the similarity of the pharmacokinetics of the two study drugs.

The investigator will perform safety evaluation for vital signs, physical examinations, ECG, clinical laboratory tests and adverse events throughout the study. Immunogenicity evaluation (ADA, ADA titration and nAb) will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy subjects aged from 18 to 50 years (including the boundary value)
* Normal vital signs, physical examinations, ECG, clinical laboratory tests and imageological examination results or abnormal with no clinical significance according to the doctor's judgment;
* Body weight between 50-90kg and BMI between 19.0-26.0kg/m2 (including boundary value);

Exclusion Criteria:

* People who have previously used or participated in clinical trials of monoclonal antibody with the same target or dupilumab
* People with a clear history of allergy and/or allergy to monoclonal antibodies of the same target /investigational drugs and their components.
* People who have special dietary requirements or are unable to follow a uniform diet.
* Dizzy blood, dizzy needle history. Blood donation > 400 ml within 3 months or > 200 ml within 4 weeks prior to screening, or planning to donate blood during the study.
* Having participated in drug or device clinical trials within 3 months or 5 half-lives of other investigational drugs before the study administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2024-08-31 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Endpoint | 0-8weeks
  Cmax
Pharmacokinetics Endpoint | 0-8weeks
  AUC0-∞

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China